CLINICAL TRIAL: NCT02463656
Title: Growth Arrest in Focal Dermal Hypoplasia
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2127
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Focal Dermal Hypoplasia
MeSH Terms: conditions — Focal Dermal Hypoplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Focal dermal hypoplasia (FDH) is a rare genetic disorder of ectodermal dysplasia caused by mutation in the Porcupine Homolog (Drosophila) (PORCN) gene which results in skin, hair, limb and eye abnormalities. Short stature and underweight have been noted in the majority of these patients. Since the pituitary gland arises from ectodermal tissue, the investigators suspect that pituitary deficiencies may contribute to poor linear growth. This study will examine the nutritional, gastrointestinal and endocrine mechanisms that may account for linear growth stunting and low weight that is observed in FDH. The investigators will utilize standard clinical tools including a bone age xray, glucagon stimulation test to evaluate growth hormone status, baseline laboratory analysis of hormone and nutritional/gastrointestinal markers, food diaries, symptom diaries, and growth charts.

DETAILED DESCRIPTION:
Focal dermal hypoplasia (FDH) is a rare genetic disorder of ectodermal dysplasia caused by mutation in the Porcupine Homolog (Drosophila) (PORCN) gene which results in skin, hair, limb and eye abnormalities. Short stature and underweight have been noted in the majority of these patients. Since the pituitary gland arises from ectodermal tissue, the investigators suspect that pituitary deficiencies may contribute to poor linear growth. This study will examine the nutritional, gastrointestinal and endocrine mechanisms that may account for linear growth stunting and low weight that is observed in FDH. The investigators will utilize standard clinical tools including a bone age xray, glucagon stimulation test to evaluate growth hormone status, baseline laboratory analysis of hormone and nutritional/gastrointestinal markers, food diaries, symptom diaries, and growth charts.

ELIGIBILITY:
Inclusion Criteria:

* patients with focal dermal hypoplasia
* between the ages of 3 and 18 years
* ability to fast overnight, and
* weight at least 9 kg

Exclusion Criteria:

* pregnant individuals,
* weight less than 9 kg

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with focal dermal hypoplasia
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Determination of Growth Hormone Deficiency | 1 day
  Glucagon growth hormone stimulation test

SECONDARY OUTCOMES:
Determination of poor growth | 1 day
  Bone age x-rays will be read independently and compared to the accepted standards and quantified as a standard deviation from chronological age.
Determination of poor weight gain | 1 day
  Evaluation of IGF-1 levels which are frequently low in children who are underweight or poorly nourished.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie C Hsu, MD, Principal Investigator — University of Colorado, Denver